CLINICAL TRIAL: NCT04132388
Title: Hidradenitis Suppurativa Patients' Experience of Treatment With Adalimumab
Brief Title: Hidradenitis Suppurativa Patient Experience With Humira Treatment
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor and site agreed the research would not happen now; several delays and other issues
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB00050544
Record Dates: First submitted 2019-09-13; First posted 2019-10-18 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Hidradenitis Suppurativa
Keywords: adalimumab; medical adherence
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: This is a prospective single-center open-label randomized 6 month study. There will not be a washout period.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized to either standard-of-care or to an electronic reporting intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard-of-Care (Active Comparator): Subjects will be instructed to take adalimumab according to the labeled dosing regimen. Subjects will return for evaluation at 12 & 26 weeks (or end of study). At each visit the subject will be scored for disease severity and adverse events. The assessor of these measures will be blinded to treatment group assignment. At the baseline and at the end of therapy visit (26 weeks), all subjects will complete a HS self-assessment questionnaire, treatment satisfaction questionnaire and physician trust survey. Pregnancy tests will be completed on females of childbearing potential at the baseline visit.
  Interventions: Drug: Adalimumab
- Electronic Reporting (Experimental): Subjects will be instructed to take adalimumab according to the labeled dosing regimen. The electronic reporting intervention consists of reporting the experience with the treatment (whether the treatment was taken, the efficacy of the treatment, and any issues that have come up) at weekly intervals for 6 weeks, then every 4 weeks thereafter.
  Subjects will return for evaluation at 12 & 26 weeks (or end of study). At each visit the subject will be scored for disease severity and adverse events. The assessor of these measures will be blinded to treatment group assignment. At the baseline and at the end of therapy visit (26 weeks), all subjects will complete a HS self-assessment questionnaire, treatment satisfaction questionnaire and physician trust survey. Pregnancy tests will be completed on females of childbearing potential at the baseline visit.
  Interventions: Other: Electronic Reporting; Drug: Adalimumab

INTERVENTIONS:
Other: Electronic Reporting — The electronic reporting intervention consists of reporting the experience with the treatment (whether the treatment was taken, the efficacy of the treatment, and any issues that have come up) at weekly intervals for 6 weeks, then every 4 weeks thereafter.
  Subjects will return for evaluation at 12 & 26 weeks (or end of study). At each visit the subject will be scored for disease severity and adverse events. The assessor of these measures will be blinded to treatment group assignment. At the baseline and at the end of therapy visit (26 weeks), all subjects will complete a HS self-assessment questionnaire, treatment satisfaction questionnaire and physician trust survey. Pregnancy tests will be completed on females of childbearing potential at the baseline visit.
  Arms: Electronic Reporting
Drug: Adalimumab — Subjects will be instructed to take Humira according to the labelled dosing regimen. Treatment will be for 26 weeks
  Other Names: Humira

SUMMARY:
Hidradenitis suppurativa (HS) is a chronic relapsing condition with significant psychosocial impact and morbidity, but that doesn't mean that patients will necessarily be adherent to recommended treatments. Patients, especially those on chronic medication therapy, inevitably miss doses. They use too little or too much therapy. They may take medications too soon or too far apart. While adherence to injection treatments tend to be better than adherence to topical or oral treatment, adherence to injections may still be poor.

Traditional methods for measuring medical adherence-including questionnaires, surveys, and diaries- tend to be unreliable overestimate adherence. Chemical markers are problematic because of the tendency for patients to use their medication right before visits, so called "white coat compliance." Our research team has pioneered the use of electronic monitoring devices which measure and record the date and time of medication events to assess adherence in dermatology. The study team have demonstrated the feasibility of using such monitors to measure adherence to adalimumab in patients with psoriasis. Although only a small study, it documented a broad range of how patients use adalimumab and found that adherence was poor in about half of the patients. While the impact of psoriasis on patients' lives is large, adherence is still poor. How adherent patients with hidradenitis are to weekly adalimumab treatment is not yet well characterized.

DETAILED DESCRIPTION:
This is a prospective single-center open-label randomized 6 month study. There will not be a washout period. Treatment will be for 26 weeks.

Subjects will have baseline disease severity assessments. Subjects will be instructed to take adalimumab according to the labelled dosing regimen. Subjects will be randomized to either standard-of-care or to an electronic reporting intervention.

The reporting intervention consists of reporting the experience with the treatment (whether the treatment was taken, the efficacy of the treatment, and any issues that have come up) at weekly intervals for 6 weeks, then every 4 weeks thereafter.

Subjects will return for evaluation at 12 & 26 weeks (or end of study). At each visit the subject will be scored for disease severity and adverse events. The assessor of these measures will be blinded to treatment group assignment. At the baseline and at the end of therapy visit (26 weeks), all subjects will complete a HS self-assessment questionnaire, treatment satisfaction questionnaire and physician trust survey. Pregnancy tests will be completed on females of childbearing potential at the baseline visit.

Primary Endpoints: Adherence to adalimumab treatment

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 18 - 70
* Diagnosis of HS for which adalimumab is indicated according to the adalimumab prescribing information.
* All subjects must have a negative TB skin test according to prescribing guidelines.
* Subjects must be starting adalimumab for the first time, prescribed by their dermatologist.

Exclusion Criteria:

* All experimental drugs or devices are to be discontinued at least 1 month prior to initiation of study therapy.
* Subjects who are receiving biologic therapy with a potential therapeutic impact on hidradenitis within 3 months will be excluded.
* Pregnant and nursing females will not be allowed in the study, and females of childbearing potential will have a pregnancy test at baseline. Females of childbearing potential must agree to use approved birth control methods for the duration of the study.
* Subjects who have received live vaccines within a 3 month period prior to enrollment will also be excluded.
* In addition, subjects who have any skin condition or disease that may require concurrent therapy or may confound the evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-20 (Estimated); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Number of days between each dose for all subjects | week 12 post randomization
  assessment of adalimumab treatment
Number of days between each dose for all subjects | week 26 post randomization
  assessment of adalimumab treatment
Percentage of patients who achieve adherence success | week 12 post randomization
  percentage who have taken over 90% of correct doses of study drug
Percentage of patients who achieve adherence success | week 26 post randomization
  percentage who have taken over 90% of correct doses of study drug

SECONDARY OUTCOMES:
Number of Doses Taken | week 12 post randomization
  Measured by MEMs cap
Number of Doses Taken | week 26 post randomization
  Measured by MEMs cap
Physician Global Assessment (PGA) | week 12 post randomization
  Assessment score ranges from 0 to 5 with a higher score denoting a worse outcome.
Physician Global Assessment (PGA) | week 26 post randomization
  Assessment score ranges from 0 to 5 with a higher score denoting a worse outcome.
Hidradentis Suppurativa Clinical Response (HiSCR) | week 12 post randomization
  Hidradenitis Suppurativa Clinical Response (HiSCR) measures number of inflammatory lesions.
Hidradentis Suppurativa Clinical Response (HiSCR) | week 26 post randomization
  Hidradenitis Suppurativa Clinical Response (HiSCR) measures number of inflammatory lesions.
Dermatology Life Quality Index (DLQI) | week 12 post randomization
  Scale ranges from 0 to 30 with a higher rating denoting a worse outcome.
Dermatology Life Quality Index (DLQI) | week 26 post randomization
  Scale ranges from 0 to 30 with a higher rating denoting a worse outcome.
Number of Doses Missed | week 26 post randomization
Total Time in Study | week 26 post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Rita O Pichardo, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No